CLINICAL TRIAL: NCT05930964
Title: Validity and Reliability of Persian Version of Low Physical Activity Questionnaire (LoPAQ)
Brief Title: Validity of Low Physical Activity Questionnaire (LoPAQ)
Status: Completed | Type: Observational
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA23ES-1-02
Record Dates: First submitted 2023-06-14; First posted 2023-07-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease; Hemodialysis Complication
Keywords: Hemodialysis; Physical Activity; Validity; Reliability; Sedentary Behaviour
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients: They will fill 3 questionnaires and will do some functional tests.

SUMMARY:
The goal of this observational study is to assess validity and reliability of Persian Version of Low Physical Activity Questionnaire. The main questions it mains to answer are:

What is the level of physical activity in hemodialysis patients? Is Persian Version of Low Physical Activity Questionnaire, Valid to assess physical activity levels of dialysis patients?

Is Persian Version of Low Physical Activity Questionnaire, reliable?

Participants will answer 3 questionnaires and will do some functional tests.

DETAILED DESCRIPTION:
Currently, between 8 and 16 percent of the world's population is suffering from chronic kidney disease, and this number is increasing day by day, and it is predicted that by 2040, kidney disease will be the fifth cause of death.

End-stage kidney disease patients, especially hemodialysis patients, face various problems, and during the years of dialysis, they suffer from many complications and problems, such as repeated hospitalizations, reduced physical performance, reduced aerobic capacity, low quality of life, and having a sedentary life. suffer, so that the activity level of these patients is between 20 and 50% of healthy people.

The physical activity level of patients undergoing hemodialysis treatment is low and significantly lower than the same inactive control groups. Research has shown that the level of physical activity of hemodialysis patients gradually decreases by approximately 4.5% per month during the entire period of the disease . In addition, the activities related to the work done at home constitute the largest part of the energy consumption of hemodialysis patients, which means that the types of activities of hemodialysis patients are usually limited to the lower category.

Valid instruments for measuring physical activity at the low end of the physical activity range and producing quantitative results are required among dialysis patients who are extremely inactive. This study aimed to translate and adapt a Persian version of the low physical activity questionnaire (LoPAQ) and to examine its reliability and validity among hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* On hemodialysis for ≥3 months
* Able to walk without assistance
* Ability to provide informed consent and complete the questionnaires

Exclusion Criteria:

* Diagnosis of mental or cognitive disorders
* Unstable conditions
* Hospitalization in the previous 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients being treated with the same respective dialysis modalities for at least 3 months and being ambulatory (with or without assistive device) will be included.
  But non-ambulatory patients having significant cognitive dysfunction, progressive degenerative,neurologic disease or severe rheumatologic or orthopedic conditions, angina upon exertion, or myocardial infarction or cardiac surgery within the last year will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Content validity of the Low Physical Activity questionnaire | Through out study completion, an average of 1 weeks
  Content validity Content validity of the questionnaire was measured using the content validity index (CVI). The item-level CVI will be calculated as the percentage of specialists giving a rating of either 3 or 4. Generally, a CVI higher than 0.78 suggest good content validity.
Physical Activity Level | Through out study completion, an average of 1 weeks
  Physical activity level was assessed by Low Physical Activity Questionnaire (LoPAQ).
Physical Activity Level | Through out study completion, an average of 1 weeks
  Physical activity level was assessed by Community Health Adults Model Program for Seniors (CHAMPS) questionnaire.
Test-retest reliability of Low Physical Activity Questionnaire (LoPAQ) | Through out study completion, an average of 2 weeks
  Test-retest reliability of Low Physical Activity Questionnaire (LoPAQ) was determined by calculating the intraclass correlation coefficient (ICC,two-way mixed analysis of variance).

SECONDARY OUTCOMES:
Self-reported physical function level | Through out study completion, an average of 1 weeks
  Self-reported physical function was assessed using the Physical Function scale of the Quality of Life questionnaire
Physical performance | Through out study completion, an average of 1 weeks
  Physical performance was assessed using the Short Physical Performance Battery test. The range of this test score is 0-12. Those who have disabilities in the activity of their daily living will take lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: MohammadAli Tabibi, PhD, Principal Investigator — Pardis Specialized Wellness Institute
Locations (1):
- Khorshid Dialysis Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data will be available after the paper is published. No end date.
Supporting Information: SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Data will be accessible with no criteria. Anyone who wishes will have access to data.

REFERENCES:
- [Result] Huang M, Lv A, Wang J, Xu N, Ma G, Zhai Z, Zhang B, Gao J, Ni C. Exercise Training and Outcomes in Hemodialysis Patients: Systematic Review and Meta-Analysis. Am J Nephrol. 2019;50(4):240-254. doi: 10.1159/000502447. Epub 2019 Aug 27. PMID 31454822
- [Result] Bao Y, Dalrymple L, Chertow GM, Kaysen GA, Johansen KL. Frailty, dialysis initiation, and mortality in end-stage renal disease. Arch Intern Med. 2012 Jul 23;172(14):1071-7. doi: 10.1001/archinternmed.2012.3020. PMID 22733312
- [Result] Johansen KL, Chertow GM, Kutner NG, Dalrymple LS, Grimes BA, Kaysen GA. Low level of self-reported physical activity in ambulatory patients new to dialysis. Kidney Int. 2010 Dec;78(11):1164-70. doi: 10.1038/ki.2010.312. Epub 2010 Sep 1. PMID 20811334
- [Result] Johansen KL, Kaysen GA, Dalrymple LS, Grimes BA, Glidden DV, Anand S, Chertow GM. Association of physical activity with survival among ambulatory patients on dialysis: the Comprehensive Dialysis Study. Clin J Am Soc Nephrol. 2013 Feb;8(2):248-53. doi: 10.2215/CJN.08560812. Epub 2012 Nov 2. PMID 23124787
- [Result] Johansen KL, Painter P, Delgado C, Doyle J. Characterization of physical activity and sitting time among patients on hemodialysis using a new physical activity instrument. J Ren Nutr. 2015 Jan;25(1):25-30. doi: 10.1053/j.jrn.2014.06.012. Epub 2014 Sep 8. PMID 25213326
- [Result] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Derived] Tabibi MA, Samouei R, Salimian N, Shahidi S, Atapour A, Nazemi F, Ghenaat M, Nikbakht S, Sarbazi MH, Soleymany M, Roshanaeian Z, Khajeheian B, Khaki Z, Sokani AS, Ebrahimi R, Ahmadi S. Validity and reliability of Persian version of Low Physical Activity Questionnaire (LoPAQ). BMC Nephrol. 2024 May 22;25(1):178. doi: 10.1186/s12882-024-03615-w. PMID 38778292